CLINICAL TRIAL: NCT05159882
Title: A Multicenter, Randomized, Double-Blind, Parallel, Active-Controlled Phase III Study on Metformin Combined With THR-1442 or Dapagliflozin in T2DM
Brief Title: Safety and Efficacy of THR-1442 Compared to Dapagliflozin as Add-on Therapy to Metformin in T2DM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newsoara Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Newsoara HYK Biopharmaceutical (Shanghai) Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THR-1442-C-606
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-11

CONDITIONS: T2DM
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: THR-1442 tablets, 20 mg; Double-Blind; Each subject will receive THR-1442, 20 mg once daily for the duration of the study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Dapagliflozin tablets, 10mg; Double Blind; Each subject will receive Dapagliflozin (active tablet) once daily for the duration of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THR-1442 20mg (Experimental): Each subject will receive THR-1442 20 mg and Dapagliflozin placebo, once daily for the duration of the study.
  Interventions: Drug: THR-1442 and Dapagliflozin placebo
- Dapagliflozin10mg (Active Comparator): Each subject will receive Dapagliflozin 10 mg and THR-1442 placebo, once daily for the duration of the study.
  Interventions: Drug: Dapagliflozin 10mg and THR1442 placebo

INTERVENTIONS:
Drug: THR-1442 and Dapagliflozin placebo — THR-1442 tablets 20mg and Dapagliflozin tablets placebo
  Arms: THR-1442 20mg
Drug: Dapagliflozin 10mg and THR1442 placebo — Dapagliflozin tablets 10mg and THR-1442 tablets placebo
  Arms: Dapagliflozin10mg

SUMMARY:
The purpose of this study is to investigate the effect of THR-1442 compared to Dapagliflozin as an add-on therapy to metformin in lowering hemoglobin A1c (HbA1c) levels in subjects with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Approximately 390 subjects with inadequately controlled T2DM on metformin were to be recruited from China. Subjects were randomly assigned to receive THR-1442 tablet, 20 mg, or Dapagliflozin tavlet,10 mg, in a ratio of 1:1 once daily for 24 weeks. Subjects were to continue taking metformin for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult subjects ≥ 18 years of age
2. If subjects are female of childbearing potential, subjects must be negative on the pregnancy test and abstain from coitus or use effective contraceptive measures during the entire study until 30 days after the investigational product is discontinued
3. Subjects diagnosed with T2DM, with a HbA1c level of 7.5-11% (inclusive) at screening and 7.0-10.5% (inclusive) at enrollment
4. Subjects who are treated with a stable dose of ≥ 1500 mg/day metformin monotherapy along with diet and exercise counseling for at least 8 weeks prior to screening
5. Subjects with a BMI of 19-35kg/m2 (inclusive) at screening
6. If applicable, taking stable doses of treatment for dyslipidemia and/or hypertension for 30 days prior to screening. Subjects who do not need to be treated with dyslipidemia or hypertension by the investigator's judgment are also eligible for the study

Exclusion Criteria:

1. History of diabetes insipidus
2. Definitive diagnosis of Type 1 diabetes mellitus, maturity-onset diabetes of the young (MODY), or secondary diabetes mellitus
3. Symptoms of diabetes mellitus inadequate control, resulting in the inability to participate in this trial, including but not limited to significant polyuria and polydipsia within 3 months prior to the screening visit and weight loss > 10%
4. History of urinary tract or genital infection within 6 months prior to screening, or ≥ 3 times of urinary tract or genital infections within 6 months prior to screening that require treatments
5. Two or more consecutive SMBG measures ≥ 250 mg/dL (13.9 mmol/L) prior to randomization (run-in period) accompanied by clinical signs or symptoms of hyperglycemia prior to randomization, including weight loss, blurred vision, increased thirst, increased urination, or fatigue
6. History of diabetic ketoacidosis or hyperosmolar non-ketonic coma within 6 months prior to screening
7. History of severe fracture secondary to osteoporosis
8. Poorly controlled hypertension: blood pressure systolic ≥ 160 mmHg and/or blood pressure diastolic ≥ 100 mmHg
9. Surgical history resulting in unstable weight or scheduled for such surgery during the study period
10. Any unstable endocrine, psychiatric, or rheumatoid disease as assessed by the investigator
11. Possible risk of dehydration or body fluid exhaustion based on the investigator's judgment that may affect the interpretation of efficacy or safety data
12. Currently having or had a history of alcohol or drug abuse within the past 6 months
13. Presence of the following cardiovascular/vascular disorders within 6 months prior to screening:
14. Unstable or rapidly progressive renal disorder
15. Congenital renal glycosuria
16. Major liver disease, including but not limited to hepatitis chronic active and/or significant hepatic function abnormal, including ALT and/or AST ≥ 3 × upper limit of normal (ULN) and/or total bilirubin ≥ 2 × ULN; or medical history of severe hepatobiliary disease; or history of any drug-related hepatotoxicity;
17. Current positive serological test result for infectious hepatitis, including known positivity to hepatitis B surface antigen and hepatitis C antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in HbA1c at Week 24 | Baseline to week 24
  HbA1c was obtained at baseline and at Week 24

SECONDARY OUTCOMES:
Change From Baseline in FPG at Week 24 | Baseline, up to 24 weeks
  FPG was obtained at baseline and at Week 24
Change in Body Weight From Baseline to Week 24 | Baseline, up to 24 weeks
  Body Weight was obtained at baseline and at week 24
Changes in blood pressure from baseline to week 24 | Baseline, up to 24 weeks
  Blood pressure was obtained at baseline and at week 24

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Shandong Province Qianfoshan Hospital, Jinan, Shandong
  - Affiliated Huzhou Hospital Zhejiang University School of Medical, Huzhou, Zhejiang
  - China-Japan Friendship Hospital, Beijing